CLINICAL TRIAL: NCT05292963
Title: Goodwill of Central Texas: Fatherhood Works Program Evaluation
Brief Title: Goodwill of Central Texas: Fatherhood Works Healthy Marriage and Responsible Fatherhood Program Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Evaluation & Research (Other)
Collaborators: Goodwill of Central Texas (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #2021/03/31
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Results first posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Fathers

STUDY DESIGN:
Intervention Model Description: Participants receive 26 hours of Nurturing Fathers curriculum, delivered in person or virtually over Zoom. Participants also receive employment supports, case management, and financial literacy training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fatherhood Works Program delivered in-person (Experimental): Participants receive 26 hours of Nurturing Fathers curriculum, delivered in person. Participants also receive employment supports, case management, and financial literacy training.
  Interventions: Other: Intervention #1: Fatherhood Works Program Delivered to Participants

INTERVENTIONS:
Other: Intervention #1: Fatherhood Works Program Delivered to Participants — Participants receive 26 hours of Nurturing Fathers curriculum, delivered in person. Participants also receive employment supports, case management, and financial literacy training.

SUMMARY:
The key goal of this descriptive evaluation is to assess the extent to which participation in the Fatherhood Works Program is positively associated with improved attitudes and behaviors among fathers and father figures in Central Texas. Research questions will focus on whether attitudes and behaviors related to parenting, co-parenting, and employment change after participation in primary program services.

DETAILED DESCRIPTION:
This evaluation seeks to understand the positive and/or negative impacts of an evidence-based core curriculum, Nurturing Fathers (NF), in combination with other workshops and case management services. All participants will receive a range of support services tailored to individuals' needs related to financial planning, career counseling, job search assistance, and occupational skills training. The program facilitator will offer the NF curriculum in both virtual and in-person formats. The evaluation will seek to determine to what extent participation in a program that uses Nurturing Fathers curriculum, in combination with other workshop programming, is associated with changes in parenting and employment attitudes as well as parenting and co-parenting behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Father figure
* Child up to 24 years of age
* Resides in Central Texas
* Adult (age 18 and older)

Exclusion Criteria:

* Minor (under the age of 18)
* Not a father/father figure
* Resides outside of Central Texas
* Child is older than 24 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2025-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matt D Shepherd, PhD, Principal Investigator — Midwest Evaluation and Research
Locations (1):
- Goodwill of Central Texas, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
All participant data will be confidential and aggregated. No individual participant data will be released unless requested by the courts. This study looks at data as a whole.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fatherhood Works Program Delivered In-person
Started | 395
Completed | 395
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fatherhood Works Program Delivered In-person
Number analyzed (Participants) | 395
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 392
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 35.6 [19 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190
  Male | 205
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 130
  Not Hispanic or Latino | 261
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 16
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 8
  Black or African American | 225
  White | 126
  More than one race | 16
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Parenting Behavior Measurement #1
Description: 1a) Will participants report significantly healthier parenting behavior after completing primary educational services and employment support services?
  Items measured include:
  1 item: frequency reaching out to children (categories, 5-point scale) 7 items: frequency engaging in key behaviors (categories, 5-point scale)
  Measured on the Healthy Parenting Behavior Scale #1 as:
  1 = never, 2 = 1 to 2 days per month, 3= 3 or 4 days per month, 4 = 2 or 3 days per week, 5 = every day or almost every day
  The 8 items are measured as a construct. All items are added together and divided by 8 to create the construct score. The higher the score, the better the outcome.
  maximum score of 5.0, minimum score of 1.0
Time Frame: Change from baseline in parenting behavior (interaction with child) from enrollment to 12-month follow-up
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Fatherhood Works Program Delivered In-person
Number analyzed (Participants) | 169
score on scale
  mean at baseline | 4.23 (.656)
  mean at follow-up | 4.34 (.629)

2. Primary Outcome: Co-parenting Behavior Measurement #1
Description: 2) Will participants report significantly healthier co-parenting behavior after completing primary educational services and employment support services?
  Items measured include:
  11 items: frequency of agreement with key co-parenting behaviors (interval, 5-point scale)
  Measured on the Healthy Co-parenting Behavior Scale #1 as:
  1 = Strongly Disagree, 2 = Disagree, 3= Neutral, 4 = Agree, 5 = Strongly Agree For 6 items, the lower the rating, the better the score. 5 items are reverse coded, with a higher rating indicating a better score.
  The 11 items are measured as a construct. All items are added together and divided by 8 to create the construct score. The higher the score, the better the outcome.
  maximum score of 5.0, minimum score of 1.0.
Time Frame: Change from baseline in co-parenting behavior (interaction with co-parent) from enrollment to 12-month follow-up
Measure: Mean (Standard Deviation); unit: scale on score
Arm/Group | Fatherhood Works Program Delivered In-person
Number analyzed (Participants) | 135
scale on score
  mean at baseline | 3.682 (.837)
  mean at follow-up | 3.64 (.818)

3. Secondary Outcome: Healthy Parenting Attitudes Measurement #1
Description: Will participants report significantly healthier parenting attitudes after completing primary educational services and employment support services?
  Items measured include:
  Parenting attitudes measured with:
  7 items - frequency of key parenting attitudes toward children (categories, 5-point scale)
  Measured on the Healthy Parenting Attitude Scale #1 as:
  1 = Always, 2 = Often, 3= Sometimes, 4 = Rarely, 5 = Never For 3 items, the lower the rating, the better the score. 4 items are reverse coded, with a higher rating indicating a better score.
  The 8 items are measured as a construct. All items are added together and divided by 8 to create the construct score. The higher the score, the better the outcome.
  maximum score of 5.0, minimum score of 1.0
Time Frame: Change from baseline in parenting attitudes (attitudes toward child) from enrollment to immediately after program completion (7 weeks).
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Fatherhood Works Program Delivered In-person
Number analyzed (Participants) | 165
score on scale
  mean at baseline | 4.52 (.430)
  mean at follow-up | 4.55 (.365)

4. Secondary Outcome: Healthy Employment Attitudes Measurement #1
Description: Items measured include:
  5 items: level of agreement with attitudes related to job searching
  Measured on the Healthy Employment Attitude Scale as:
  1 = Strongly Disagree, 2 = Disagree, 3= Neutral, 4 = Agree, 5 = Strongly Agree
  The 5 items are measured as a construct. All items are added together and divided by 5 to create the construct score. The higher the score, the better the outcome.
  maximum score of 5.0, minimum score of 1.0.
Time Frame: Time frame: Change from baseline in co-parenting behavior (interaction with co-parent) from enrollment to 12-month follow-up.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Fatherhood Works Program Delivered In-person
Number analyzed (Participants) | 173
score on scale
  mean at baseline | 4.42 (.771)
  mean at follow-up | 4.42 (.683)

ADVERSE EVENTS:
Time Frame: 1 year through study completion
Description: The definitions of adverse events do not differ from the clinicaltrials.gov definitions.
Arm/Group | Fatherhood Works Program Delivered In-person
All-Cause Mortality (participants affected / at risk) | 0/395
Serious Adverse Events (participants affected / at risk) | 0/395
Other Adverse Events (participants affected / at risk) | 0/395

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2025-01-09): https://cdn.clinicaltrials.gov/large-docs/63/NCT05292963/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-09): https://cdn.clinicaltrials.gov/large-docs/63/NCT05292963/SAP_001.pdf